CLINICAL TRIAL: NCT02636881
Title: Focal Cartilage Defects in the Knee -A Randomized Controlled Trial Comparing Autologous Chondrocyte Implantation With Arthroscopic Debridement
Brief Title: Autologous Cartilage Implantation vs Arthroscopic Debridement
Acronym: ACI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Asbjorn Aroen, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/2200
Record Dates: First submitted 2015-12-14; First posted 2015-12-22 (Estimated); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Knee Injury; Cartilage Injury
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous Chondrocyte Implantation (Active Comparator): A diagnostic arthroscopy of the knee joint.The lesion is stabilized down to the subchondral bone, but not through it. Cartilage biopsy is taken from the medial femoral notch. The harvested cartilage is transported to the cell culture Laboratory and cultured for two weeks. The chondrocyte implantation: A mini-open arthrotomy is performed and the lesion is curetted down to subchondral bone, avoiding bleeding. The lesion is measured and a template of sterile aluminum foil is used to cut out a matching piece of collagen sheet which is used to contain the cells in the defect. The flap is sutured to the lesion and sealed with fibrin glue, leaving and opening at the upper part for injection of the cells. The last opening is then closed with a last stitch and fibrin glue.
  Interventions: Procedure: Autologous Chondrocyte Implantation
- Arthroscopic Debridement (Sham Comparator): The AD group will be subjected to a diagnostic arthroscopy with a full inspection of the knee joint to ensure the inclusion criteria are fulfilled. Lose bodies are removed, any meniscal pathology is addressed. Inflamed synovium is debrided. The lesion is stabilized by debridement around the edges and down to the subchondral bone using a ring curette, but not through it. Microfracture or any other cartilage treatment will not be performed.
  No intra-articular local anesthetics will be used due to the possible harmful effect on cartilage [41-43].
  All the operating surgeons will receive proper training in the operative procedure before study start.
  Interventions: Procedure: Arthroscopic Debridement

INTERVENTIONS:
Procedure: Autologous Chondrocyte Implantation — Implantation of the patients own cartilage cells in a chondral defect of the knee
  Arms: Autologous Chondrocyte Implantation
Procedure: Arthroscopic Debridement — Arthroscopic diagnosis and debridement of the lesion, without cartilage therapy. Removal of lose bodies etc.
  Arms: Arthroscopic Debridement

SUMMARY:
82 patients aged 18-49 years with an isolated focal cartilage defect in the knee will be randomized to either receive autologous cartilage implantation or arthroscopic debridement. Both groups will then undergo a systematic physiotherapy training regime for 6-9 months. The Groups will then be compared for results, after 3, 6, 12 and 24 months, by using validated patient reported outcome scores (Lysholm, KOOS, Tegner) and EQ5D (European Quality of Life 5 dimensions) as well as clinical examination and radiological findings at 2 years (MRI).

DETAILED DESCRIPTION:
Details Focal cartilage defects in the knee - A randomized controlled trial comparing Autologous Chondrocyte Implantation with arthroscopic debridement Clinical Compare the effect of Autologous Chondrocyte Implantation (ACI) with arthroscopic debridement (AD) in patients with symptomatic full thickness knee cartilage injuries larger than 2cm2.

Focal cartilage injuries in the knee might have devastating effect both in the short term and in the long term. Various surgical treatment options are available; with ACI established as a recognized treatment method for larger lesions. Meta-analysis and systematic reviews have required well-designed, long-term, multicenter studies to evaluate clinical outcomes of ACI with the use of a "no treatment" group as a control group.

H0: There is no difference in KOOS QoL after ACI or AD from baseline to 24 months after surgery.

H1: There is a difference in KOOS QoL after ACI or AD from baseline to 24 months after surgery.

Questionnaires: KOOS, Tegner score, Lysholm score, EQ-5D, VAS (Visual analogue scale).

Physical examination: range of motion and hop test. Radiology: x-ray and MRI of the knee. Primary aim: KOOS quality of life (QoL) subscore. Prospective, single-blinded parallel-group bicenter study with 2 treatment arms.

Approx. 36 months inclusion and 24 months follow up. In total 5 years. 24 months. All will be invited to participate in late controls after 5 and 10 years.

2 Norwegian hospitals: Akershus University Hospital and Oslo University Hospital - Ullevål.

82 patients Inclusion: age 18-50 years old, single symptomatic cartilage defect on femoral condyle or trochlea, defect size larger than 2 cm2, defect ICRS (International Cartilage Repair Society) grade 3-4, ligamentous stable knee, range of motion 5-105°, Lysholm score < 75 and informed consent.

Exclusion: Osteoarthritis, rheumatoid or other systemic arthritis, malalignment > 5° measured on x-rays, BMI > 30, comorbidities that may influence surgery or rehabilitation, pregnancy, inability to complete questionnaires or rehabilitation, serious alcohol or drug abuse, previous cartilage surgery to the chondral defect except OCD (osteochondritis dissecans)surgery.

2 treatment groups with 41 patients in each group. 3 months (± 2 weeks), 6 months (± 4 weeks), 12 months (± 6 weeks) and 24 months (± 8 weeks). All will be invited to participate in late controls after 5 and 10 years.

If any unforeseen complication outside normal clinical practice occurs, the sponsor representative will be contacted as soon as possible with a parallel message to the local coordinators at the involved hospitals. During each follow up, there will be a case report form (CRF) regarding complications and safety.

A 5 mL venous blood sample will be drawn on the day of operation. The blood sample will be centrifuged before serum is pipetted in a sterile tube. The serum will be analyzed at Oslo University Hospital - Rikshospitalet on the cartilage biomarker microRNA-140 (miR-140).

During the open chondrocyte implantation the excess cartilage debrided from the rim of the lesion will be sent for similar microRNA-140 (miR-140) analysis. (applicable for the 41 patients in the ACI arm only) If normal distribution, aims will be analyzed using linear mixed models (LMM), and the primary aim will be performed as a post hoc test for the LMM, similar to performing a two-sample t-test. If no normal distribution, analysis will be performed using Mann-Whitney U-test.

Detecting a difference of 10 in primary aim with 80% power using a standard deviation of 15. A p < 0,05 is statistically significant. This gives 37 patients in each group, adding 10% drop out meaning 41 patients in each group and 82 in total.

No interim analysis will be done. Monitor at Akershus University Hospital. Inclusion of 82 patients. The end of this study is 24 months after the last included patient. Inability to include 82 patients in 3 years. May prolong the inclusion period, or add other including hospitals in the study.

ELIGIBILITY:
Inclusion Criteria:

* Single symptomatic lesion of the trochlea, medial or lateral femoral condyle of the knee larger than 2 cm2.
* Cartilage lesion ICRS grade 3 or 4.
* More than 50 % of the menisci intact.
* Ligamentous stable knee
* Lysholm Score < 75
* Acceptable range of motion (5-105 degrees)

Exclusion Criteria:

* Osteoarthritis
* Malalignment > 5 degrees measured on HKA (hip-knee-ankle) radiographs
* Systemic arthritis
* Previous cartilage surgery
* Obesity BMI > 30
* Serious drig or alcohol abuse
* Inability to answer questionnaires or partake in rehabilitation
* Comorbidity that may influence surgery or rehabilitation

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life | up to 24 months
  The KOOS is a validated patient oriented outcome measure validated to use in cartilage Research. It assesses five domains, and the Fifth domain (knee related quality of life) will be the primary endpoint in this study.

SECONDARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score (KOOS) Other domains | preop, 3, 6, 12 and 24 months.
  The other four domains of the KOOS score (pain, symptoms, Activity of daily living, sport and recreational function) will act as secondary endpoints
Tegner Score | preop, 3, 6, 12 and 24 months.
  A validated knee-score to assess the Level of physical activity
Lysholm Knee Score | preop, 3, 6, 12 and 24 months.
  A condition specific knee score that assesses 8 domains: limp, locking, swelling, pain, stair climbing, use of support, instability and squatting
EQ5D | preop, 3, 6, 12 and 24 months.
  A generic measure of health status that produces a simple descriptive profile of Health status used in clinical evaluation of Health care.
Visual Analogue Scale | preop, 3, 6, 12 and 24 months.
  VAS scale for pain from 0 to 10
Range of motion | preop, 3, 6, 12 and 24 months.
  Clinical evaluation of the joint range of motion
Magnetic Resonance Imaging | 24 months
  A radiographic evaluation of the cartilage injury at 2 years
A Hop test | 24 months
  Clinical evaluation of the knees agility, validated in knee sport medicine Research.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Hanvold, PT, Principal Investigator — Research coordinator; asbjørn Årøen, MD, PhD, Study Chair — Akerhus University hospital
Locations (1):
- Akershus University Hospital, Lørenskog, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No
At publication.

REFERENCES:
- [Result] Randsborg PH, Brinchmann JE, Owesen C, Engebretsen L, Birkenes T, Hanvold HA, Benth JS, Aroen A. Autologous Chondrocyte Implantation Is Not Better Than Arthroscopic Debridement for the Treatment of Symptomatic Cartilage Lesions of the Knee: Two-Year Results From a Randomized-Controlled Trial. Arthrosc Sports Med Rehabil. 2024 Feb 16;6(2):100909. doi: 10.1016/j.asmr.2024.100909. eCollection 2024 Apr. PMID 38495635
- [Derived] Banitalebi H, Owesen C, Aroen A, Tran HT, Myklebust TA, Randsborg PH. Is T2 mapping reliable in evaluation of native and repair cartilage tissue of the knee? J Exp Orthop. 2021 Apr 28;8(1):34. doi: 10.1186/s40634-021-00350-1. PMID 33913035
- [Derived] Randsborg PH, Brinchmann J, Loken S, Hanvold HA, Aae TF, Aroen A. Focal cartilage defects in the knee - a randomized controlled trial comparing autologous chondrocyte implantation with arthroscopic debridement. BMC Musculoskelet Disord. 2016 Mar 8;17:117. doi: 10.1186/s12891-016-0969-z. PMID 26956476

DOCUMENTS (1):
  • Study Protocol (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT02636881/Prot_000.pdf